CLINICAL TRIAL: NCT01262703
Title: Pilot Study of the ReZolve™ Sirolimus-Eluting Bioresorbable Coronary Stent
Brief Title: Safety Study of a Bioresorbable Coronary Stent
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REVA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCT1000
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Cardiovascular Disease
MeSH Terms: conditions — Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- REVA Medical ReZolve Stent (Experimental): ReZolve Sirolimus-Eluting Bioresorbable Coronary Stent
  Interventions: Device: ReZolve Stent

INTERVENTIONS:
Device: ReZolve Stent — ReZolve Sirolimus-Eluting Bioresorbable Coronary Stent

SUMMARY:
To evaluate the safety of a new bioresorbable (non-permanent) stent platform in native coronary arteries.

DETAILED DESCRIPTION:
Today, coronary artery disease is often treated by placing a metal stent inside the vessel that serves as a permanent scaffold. However, it is hypothesized that the stent is no longer needed once the artery has healed. This study will evaluate the safety of a bioresorbable (non-permanent) stent for the treatment of coronary artery disease. The stent is designed to restore blood flow to the artery which allows the artery to remodel (heal), and then resorb from the body. The stent supports the vessel during the critical 90-day healing process, and then gradually resorbs and is cleared from the body.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of myocardial ischemia or a positive functional study.
* Normal CK-MB.
* Target lesion must be located in a native coronary artery where target vessel diameter is ≥ 2.9 mm and ≤ 3.3 mm and target lesion length is ≤ 12 mm, both assessed by on-line QCA and IVUS
* Target lesion must be in a major artery or branch with a visually estimated stenosis of ≥ 50% and < 100% with a TIMI flow of ≥ 2.
* Staged procedures are allowed in non-target vessels >24 hours before or > 30 days after REVA stent implantation

Exclusion Criteria:

* A myocardial infarction (CK-MB or Troponin > 3 times normal) within 72 hours of the procedure, has signs or symptoms of an ongoing myocardial infarction or has any visible thrombus
* Unprotected left main coronary disease with >50% stenosis
* The target vessel is totally occluded (TIMI Flow 0 to 1)
* Target lesion involves a bifurcation (a lesion with a side branch >2.0 mm in diameter containing a >50% stenosis)
* Target lesion is located within a segment supplied by distal graft
* Target lesion has possible or definite thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Ischemia-driven Target Lesion Revascularization (TLR) | 6 months
  Defined as any clinically-driven (as defined for TLR) repeat percutaneous intervention of the target vessel or bypass surgery of the target vessel.

SECONDARY OUTCOMES:
QCA & IVUS derived parameters | 12 months
  Late Loss, Restenosis Rate, %DS, MLD & Neointimal Volume
Major Adverse Coronary Events | 60 months
  Major Adverse Cardiac Events - Combined events consisting of death, Myocardial Infarction (Q-Wave, Non Q-wave: CPK > 2xULN + MB>ULN) (MI), and target vessel revascularization (TVR).
Procedural and Technical Success | Acute
  percentage of patients with angiographic success successful delivery and deployment of the device

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil